CLINICAL TRIAL: NCT04358809
Title: A Randomized, Double-blind, Two Arm, Controlled Clinical Trial to Compare the Efficacy and Safety of Mycobacterium w (Mw) Administered Along With Standard of Care Versus Placebo Administered Along With Standard of Care, in Adult, COVID 19 Positive Patients Hospitalized But Not Critically Ill.
Brief Title: Clinical Trial of Mycobacterium w in COVID-19 Positive Patients, Hospitalized But Not Critically Ill
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cadila Pharnmaceuticals (Industry)
Collaborators: Council of Scientific and Industrial Research, India (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRSC20006
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: A randomized, double-blinded, two arms, placebo controlled, clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suspension of Mw + Standard therapy of COVID-19 (Experimental): 0.3 ml (0.1ml x 3 Injection) of intradermal Mw for 3 consecutive days + Standard therapy of COVID-19
  Interventions: Drug: Suspension of heat killed (autoclaved) Mycobacterium w
- Placebo (Placebo Comparator): 0.3 ml (0.1ml x 3 Injection) of intradermal Placebo for 3 consecutive days + Standard therapy of COVID-19
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Suspension of heat killed (autoclaved) Mycobacterium w — Suspension of heat killed (autoclaved) Mw along with Standard of care (SOC) treatment for COVID-19
  Arms: Suspension of Mw + Standard therapy of COVID-19
Other: Placebo — Placebo along with Standard of care (SOC) treatment for COVID-19
  Arms: Placebo

SUMMARY:
This is a randomized, double blind, two arms, placebo controlled, clinical trial to study to evaluate the the safety and efficacy of Mycobacterium w in combination with standard of care versus placebo with standard of care for preventing the progression of COVID-19 disease and for reduction in transfer to ICU in COVID-19 infected patients admitted to the hospital.

DETAILED DESCRIPTION:
Total 480 hospitalized adult eligible patients will be randomized in 1:1 ratio to receive either Mw+SOC or placebo+SOC for first 3 days post-randomization.

Daily clinical evaluation of patient will be performed till discharge from hospital or till ICU admission.

Study duration for each patient will be approximately up to 28 days, or discharge from hospital or transfer to ICU, whichever is earlier.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 positive patients with ordinal scale score of 3.
* Patients of either gender, age ≥ 18 years at the time of enrollment.
* Female patients who are currently using reliable methods of contraception (barrier methods and intrauterine contraceptive device), with a negative urine pregnancy test during screening and agree to informed compliance of contraceptive method until at least 3 months post-dosing.
* The patients must be able and willing to comply with the study protocol, available and willing to complete all the study assessments and must have signed an Informed Consent Form.

Exclusion Criteria:

* Patient with ordinal scale of ≥4 at the time of hospital admission and randomization.
* Pregnant and / or lactating female patients.
* A family history of congenital or hereditary immunodeficiency.
* Any disease condition requiring ICU admission.
* History of dialysis, silicosis, solid organ transplantation such as renal or cardiac transplants, and disorders of the heart, or nervous system, or other metabolic inflammatory conditions, psychiatric, occupational problems that make it unlikely that the patients will comply with the protocol as determined by the investigator.
* History of administration of any immunoglobulins, any immunotherapy (antineoplastic chemotherapy, radiation therapy, immunosuppressants to induce tolerance to transplants, and corticosteroids use) and/or any blood products within the 3 months preceding study dosing, or planned future administrations during the study period.
* History of allergic reactions or anaphylaxis to Mw or its component.
* Presence of any severe systemic/autoimmune disorders as determined by medical history and/or physical examination at the time of screening, which in the judgment of the Investigator would compromise the patient's health or is likely to result nonconformance to the protocol or a patient's ability to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with increased disease severity | From baseline to Day 3, Day 7, Day 14, Day 21, Day 28 or at any time during the study till 28 days post first dosing.
  To compare the difference in proportion of patients with increased disease severity

SECONDARY OUTCOMES:
Incidence of adverse events and serious adverse events (Safety) | Till day 28
  To evaluate safety of Mw in COVID-19 patients admitted to hospital
Number of COVID-19 patients discharged from hospital | From baseline to Day 3, Day 7, Day 14, Day 21, Day 28 or at any time during the study till 28 days post first dosing.
  To compare the proportion of patients discharged from hospital
Number of COVID-19 patients transfer to ICU | From baseline to Day 3, Day 7, Day 14, Day 21, Day 28 or at any time during the study till 28 days post first dosing.
  To compare the proportion of patients transfer to ICU
Number of COVID-19 patients with reduction in disease severity by 1 ordinal scale | From baseline to Day 3, Day 7, Day 14, Day 21, Day 28 or at any time during the study till 28 days post first dosing.
  To compare the proportion of patients with reduction in disease severity by 1 ordinal scale
Number of of symptom free patients | From baseline to Day 3, Day 7, Day 14, Day 21, Day 28 or at any time during the study till 28 days post first dosing.
  To compare the proportion of symptom free patients

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Patel, MBBS, Study Chair — Cadila Pharmaceuticals Limited
Locations (4):
- India (4):
  - All India Institute of Medical Science, Raipur, Raipur, Chhattisgarh
  - All India Institute of Medical Sciences, Bhopal, Bhopal
  - Post Graduate Institute of Medical Education and Research, Chandigarh
  - All India Institute of Medical Sciences, Delhi, Delhi

IPD SHARING:
Plan to Share IPD: No